CLINICAL TRIAL: NCT05216510
Title: A Dose Finding Study for the Assessment of Delayed-type Hypersensitivity Reactions to SARS-CoV-2 Peptide Antigens in Uninfected Healthy Subjects, COVID-19 Convalescent Subjects, and COVID-19 Vaccinated Subjects
Brief Title: Assessment of Delayed-type Hypersensitivity Reactions to SARS-CoV-2 Peptide Antigens
Acronym: COVID-19 DTH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CA-C201
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Detection of Delayed-type Hypersensitivity Reactions to SARS-CoV-2 in Individuals Exposed to SARS-CoV-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Healthy uninfected/unexposed subjects to SARS-CoV-2
  Interventions: Biological: TNX-2110; Biological: TNX-2120; Biological: TNX-2130; Biological: CANDIN; Biological: Diluent
- Cohort 2 (Active Comparator): Subjects who have recovered from SARS-CoV-2 infection
  Interventions: Biological: TNX-2110; Biological: TNX-2120; Biological: TNX-2130; Biological: CANDIN; Biological: Diluent
- Cohort 3 (Sham Comparator): Subjects who have received a complete SARS-CoV-2 vaccine course
  Interventions: Biological: TNX-2110; Biological: TNX-2120; Biological: TNX-2130; Biological: CANDIN; Biological: Diluent

INTERVENTIONS:
Biological: TNX-2110 — TNX-2110 represents epitopes of multiple proteins from SARS-CoV-2 and is administered intradermally.
Biological: TNX-2120 — TNX-2120 represents the spike protein and is administered intradermally.
Biological: TNX-2130 — TNX-2130 represents non-spike proteins and is administered intradermally.
Biological: CANDIN — Candida albicans antigens to be administered intradermally as a positive control.
Biological: Diluent — Diluent consists of phosphate buffer, polysorbate 20 and mannitol and will be administered intradermally as a negative control.

SUMMARY:
This dose finding, multi-cohort study is designed to evaluate the safety and efficacy of intradermally-injectedTNX-2100, synthesized SARS-CoV-2 peptide antigens and assess the presence and magnitude of DTH reactions.

DETAILED DESCRIPTION:
Three IPs (TNX-2110, TNX- 2120, TNX-2130) will be administered by intradermal injection (0.1 mL) in two concentration strengths (Stage 1: "1:10 dilution" and Stage 2: "undiluted"). Subjects will also receive one intradermal injection (0.1 mL) of a positive control (CANDIN®), and one intradermal injection (0.1 mL) of a negative control "diluent".

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects aged 18 - 65 years of age, inclusive, in good general health as determined by medical evaluation Subject receives a negativeSARS-CoV-2 PCR test result at their screening or baseline visit

Exclusion Criteria:

Subjects will be excluded if they have clinically significant underlying conditions associated with high risk for severe COVID-19 infections as identified by the Centers for Disease Control and Prevention (CDC) (Appendix 2). These conditions include, but are not limited to: chronic obstructive pulmonary disease, diabetes mellitus (Type 1 and 2), obesity, hypertension, heart disease, and cerebrovascular disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herb Harris, MD, Study Director — Tonix Pharmaceuticals
Locations (1):
- Clinical Site, Berlin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Based on medical history, patients were assigned into 1 of the 3 groups: Cohort 1 included healthy uninfected/unexposed subject; Cohort 2 included subjects who recovered from SARS-CoV-2 infection at least 2 months prior to enrollment into the study independent of vaccination status; Cohort 3 included subjects who received a complete SARS-CoV-2 vaccine course at least 4 weeks prior to enrollment into the study with no known history of natural infection.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 1 | 1 | 7
Completed | 0 | 1 | 7
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 1 | 1 | 7 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 | 21 | 31.3 (17.45) | 29.3 (15.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 0 | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 0 | 1 | 6 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Delayed-type Hypersensitivity Reactions
Description: The primary efficacy endpoint of this study is the maximal area of induration ≥5 mm at injection sites on the volar aspect of the forearms of 3 time points post skin test administration. The outcome measure is the maximum of the area of induration of 48 hours, 72 hours, and 96 hours.
Time Frame: Up to 96 hours post skin test administration
Population: mITT Population includes all randomized subjects who completed Stages 1 and 2 of administration and had induration responses for at least one post skin test administration visit at hour 48, 72, or 96.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 1 | 1 | 6
mm | NA (NA) — Induration (Delayed-type Hypersensitivity Reactions to SARS-CoV-2 Peptide Antigens reaction) was not observed and could not be measured. | NA (NA) — Induration (Delayed-type Hypersensitivity Reactions to SARS-CoV-2 Peptide Antigens reaction) was not observed and could not be measured. | NA (NA) — Induration (Delayed-type Hypersensitivity Reactions to SARS-CoV-2 Peptide Antigens reaction) was not observed and could not be measured.

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Cohort 1: uninfected/unexposed healthy individuals
- Cohort 2: individuals confirmed to have recovered from SARS-CoV-2 infection independent of vaccination status
- Cohort 3: individuals who had received a complete SARS-CoV-2 vaccine course with no known history of natural infection
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/7
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=1) | Cohort 2 (N=1) | Cohort 3 (N=7)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 7 (7)
Swelling (General disorders) | 1 (1) | 1 (1) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all study investigators.

DOCUMENTS (2):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT05216510/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT05216510/SAP_001.pdf